CLINICAL TRIAL: NCT04786873
Title: Multicenter, Open Label Trial to Investigate the Efficacy and Safety of a Single Oral Dose of 1.0 mg/kg Macimorelin Acetate as Growth Hormone Stimulation Test (GHST) in Pediatric Patients With Suspected Growth Hormone Deficiency (GHD)
Brief Title: A Research Study of How Well Macimorelin Works to Find Out if Children Have a Lack of Growth Hormone and How Safe it is
Acronym: DETECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: AEZS-130-P02; 2018-001989-42 (EudraCT Number); U1111-1248-5075 (Other: Universal Trial Number)
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Growth Hormone Deficiency
Keywords: childhood-onset growth hormone deficiency; diagnosis of growth hormone deficiency; diagnosis of childhood-onset growth hormone deficiency; diagnostic test for growth hormone deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — macimorelin; Citrullination

STUDY DESIGN:
Intervention Model Description: This is an open label, single-dose trial to determine the diagnostic efficacy and safety of macimorelin in pediatric subjects aged 2 to less than 18 years of age in whom, based on auxological and clinical criteria, growth hormone stimulation test (GHST) is indicated due to suspected growth hormone deficiency. Four GHSTs will be conducted during the trial: the macimorelin GHST will be performed twice, and arginine and clonidine standard GHSTs will be performed once each. The macimorelin GHST will be administered at the beginning of the trial and after serial performance of the two different standard GHSTs. The macimorelin GHSTs will be performed twice to show repeatability of the macimorelin GHST. All subjects will be randomized 1:1 to the order of the arginine and clonidine GHSTs, and in a crossover manner all subjects will receive both these GHSTs.
Who Masked: Outcomes Assessor
Masking Description: This study is open label. Masking is performed with regard to the GHST results (i.e. growth hormone (GH) values).
  GH values from all GHSTs will be assessed centrally by a central lab: GH values following the two standard GHSTs at V3 and V4 will not be disclosed to the trial site prior to the end of V5 (i.e., the second macimorelin GHST). To avoid bias in the final diagnostic assessments by the investigators, macimorelin pharmacodynamic (PD) data will remain blinded to the trial sites, clinical research associates (CRAs), and trial management at contract research organization (CRO) and Sponsor until trial closure.
  An Independent Adjudication Committee (IAC) is established to perform ongoing blinded adjudication of subjects' growth hormone deficiency status. The IAC will adjudicate in a consistent manner by use of pre-defined definitions and guidelines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- standard GHST order randomized: arginine - clonidine (Active Comparator): At visit 2 (V2), all subjects will perform the macimorelin GHST and will be randomized 1:1 to the order of the clonidine and arginine GHSTs at visit 3 (V3) and visit 4 (V4).
  In this arm, those subjects will be presented which will have been randomized to the arginine GHST at V3 and the clonidine GHST at V4.
  At visit 5 (V5) all subjects will perform the macimorelin GHST.
  Interventions: Drug: Macimorelin; Diagnostic Test: Arginine; Diagnostic Test: Clonidine
- standard GHST order randomized: clonidine - arginine (Active Comparator): At V2, all subjects will perform the macimorelin GHST and will be randomized 1:1 to the order of the clonidine and arginine GHSTs at V3 and V4.
  In this arm, those subjects will be presented which will have been randomized to the clonidine GHST at V3 and to the arginine GHST at V4.
  At V5 all subjects will perform the macimorelin GHST.
  Interventions: Drug: Macimorelin; Diagnostic Test: Arginine; Diagnostic Test: Clonidine

INTERVENTIONS:
Drug: Macimorelin — Dosage form: granules for oral solution, Dosage: 1.0 mg/kg body weight, Frequency and duration: single oral dose administration. Macimorelin will be supplied in single-use aluminum pouches (synonymous: sachets) each containing 63.6 mg macimorelin as acetate, which provide 0.5 mg/mL of macimorelin when dissolved in 120 mL of water. The excess amount of 3.6 mg represents an overfill, which is needed to obtain the target concentration.
  Other Names: Macrilen; AEZS-130; Macimorelin GHST; Macimorelin test; Macrilen GHST; Macrilen test
Diagnostic Test: Arginine — For the arginine GHST, R-Gene® 10 from Pfizer will be provided as labelled investigational medicinal product (IMP). After an overnight fast, soluble arginine hydrochloride (0.5 g/kg) will be given i.v. as an infusion with an infusion duration of 30 min.
  Other Names: R-Gene 10; arginine test; arginine GHST
Diagnostic Test: Clonidine — For the clonidine GHST, CATAPRESAN® 75 tablets (Boehringer Ingelheim) will be provided as labelled IMP. Each tablet contains 75 ug clonidine hydrochloride. The tablets will be provided in boxes containing 10 tablets. The target dose is 0.15 mg/m2 body surface with a dose range of 0.08 - 0.15 mg/m2. Maximum dose will be 0.25 mg.
  After an overnight fast, clonidine (0.15 mg/m2 body surface) will be given orally.
  Other Names: Catapressan 75; Clonidine test; Clonidine GHST

SUMMARY:
This research study will find out if a new growth hormone stimulation test is safe and works as well as other tests to diagnose growth hormone deficiency (GHD) in children. The stimulation test will use a new growth hormone stimulating substance called macimorelin. By now, only adults in the USA can get this new stimulation test. The results of this study are expected to help children and teenagers with suspected GHD to get the macimorelin stimulation test.

The macimorelin test will be compared to a clonidine and an arginine test. Both are known standard stimulation tests. Altogether two macimorelin tests are planned to be performed in the study, to show how repeatable macimorelin tests results are (under a set of similar conditions).

DETAILED DESCRIPTION:
Each study participant (patient) will have 5 to 6 visits in total with the study doctor.

The study will last for about 1 to 4 months, dependent on how close the visits are done. At the visits 2, 3, 4 and 5, the patient will get a stimulation test done and blood samples will be taken. At those 4 visits, the patient will have either to drink a macimorelin drink, take some clonidine tablets or get an arginine infusion. In total, the patient will get 2 macimorelin, 1 clonidine and 1 arginine test done. The level of growth hormone (GH) will be measured 4 times during the clonidine and during the arginine test and 5 times during the macimorelin test. After the test, questions on the test tolerability will be captured from patients and parents. After the arginine test, a urine dipstick test is to be done by the patient at home.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent of subject, parent(s) or legally acceptable representative (LAR) of subject and child assent, if appropriate, must be obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
2. Male and female pediatric subjects from 2 to less than 18 years of age at the time of signing informed consent.
3. Indication for the performance of growth hormone stimulation test.
4. Presence of a height measurement minimum 6 and maximum 18 months prior to screening.

Exclusion Criteria:

1. Established diagnosis of a disease that is sufficient to explain growth deficiency or metabolic disorders that are also associated with short stature (e.g., Turner syndrome, skeletal dysplasia's, celiac disease, etc.).
2. Ongoing growth hormone therapy.
3. Presence of hypothyroidism and/or adrenal insufficiency without adequate and stable replacement therapy treatment for at least 30 days prior to first GHST.
4. Treatment with drugs directly affecting the pituitary secretion of somatotropin (e.g., somatostatin analogues, clonidine, levodopa and dopamine agonists) or provoking the release of somatostatin (antimuscarinic agents e.g., atropine).
5. Medical history of ongoing clinically symptomatic psychiatric disorders.
6. 2nd or 3rd degree atrioventricular-block, prolongation of the QRS complex over 120 milliseconds, prolongation of the QTc interval over 450 milliseconds, or any other clinically significant abnormal electrocardiogram results at the V2 pre-dose electrocardiogram (ECG) as judged by the investigator.
7. Previous participation in this trial. Participation is defined as signed informed consent.
8. Participation in any clinical trial of an approved or non-approved investigational medicinal product within 30 days before screening.
9. Known or suspected hypersensitivity to trial product(s) or related products;
10. Any disorder, which in the investigator's opinion might jeopardize subject's safety or compliance with the protocol.
11. Concomitant treatment with any drugs that might prolong QT/QTc Note: A subject who receives such treatment will not be a candidate for this study, if his/her condition does not allow for a treatment-free period of at least 5 elimination half-lives of the drug that might prolong QT/QTc before the GHST;
12. Elevation of laboratory parameters indicating hepatic or renal dysfunction or damage (aspartate amino transferase (AST), alkaline phosphatase (ALT), gamma-glutamyl transferase (GGT) > 2.5 x upper limit of normal (ULN); creatinine or bilirubin > 1.5x ULN);
13. Current active malignancy other than non-melanoma skin cancer;
14. Female of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measures as required by local regulation or practice).
15. Male of reproductive age who or whose partner(s) is not using an adequate contraceptive method (adequate contraceptive measures as required by local regulation or practice).
16. Lack of ability or willingness to give informed consent by the subject and/or his/her legal representative;
17. Anticipated non-availability for trial visits/procedures.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Area under the Receiver Operator Characteristic curve (ROC AUC) based on GH concentration during GHST following macimorelin administration | Derived from Cmax GH measurements collected in the time frame from 0 to 90 minutes after initial macimorelin GHST (visit 2 (day 0)) and GH adjudication status performed by the adjudication committee after visit 4 (between day 11 and day 58)).
  Assuming the outcome of GHD status adjudication final clinical diagnosis as the "true" GHD status, the diagnostic efficacy (estimated sensitivity, specificity, misclassification) of the macimorelin GHST will be based on the area under the receiver operating characteristic curve (ROC AUC).

SECONDARY OUTCOMES:
Sensitivity for the macimorelin GHST | Derived from Cmax GH measurements collected in the time frame from 0 to 90 minutes after initial macimorelin GHST (visit 2 (day 0)) and GH adjudication status performed by the adjudication committee after visit 4 (between day 11 and day 58)).
  Sensitivity (confirmatory secondary endpoint) will be derived from the empirical ROC plot using this GH cut-off point.
Specificity for the macimorelin GHST | Derived from Cmax GH measurements collected in the time frame from 0 to 90 minutes after initial macimorelin GHST (visit 2 (day 0)) and GH adjudication status performed by the adjudication committee after visit 4 (between day 11 and day 58)).
  Specificity (confirmatory secondary endpoint) will be derived from the empirical ROC plot using this GH cut-off point.
Overall agreement between the outcome of the macimorelin GHST and the combined outcome from the 2 standard GHSTs | Visit 4 (between day 11 and day 58)
  Agreement between the outcome of macimorelin and the combined outcome of the 2 standard GHSTs will be evaluated by 'percent overall agreement'.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola K Ammer, MD, Study Director — AEterna Zentaris
Locations (45):
- United States (12):
  - Angel Wing Clinic For Children With Diabetes, Tucson, Arizona
  - Pediatric Endocrine Associates, p.c., Greenwood Village, Colorado
  - John Hopkins All Children's Hospital, St. Petersburg, Florida
  - Emory Healthcare-Children's Center, Atlanta, Georgia
  - St. Luke's Children's Endocrinology, Boise, Idaho
  - University of Minnesota, Masonic Children's Hospital, Minneapolis, Minnesota
  - The Children's Mercy Hospital - Broadway, Kansas City, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - UNC Hospitals, Chapel Hill, North Carolina
  - Alchemi Research Center, Rosharon, Texas
  - Multicare Health System, Tacoma, Washington
- Yerevan State Medical University after Mkhitar Heraci, Yerevan, Armenia
- Georgia (3):
  - JSC Maritime Hospital, Batumi
  - National Institute of Endocrinology, Tbilisi
  - TSMU Givi Jvania Pediatric Academic Clinik, Tbilisi
- Evangelisches Klinikum Bethel, Bielefeld, Germany
- Italy (5):
  - Ospedale Pediatrico G. Salesi, Ancona
  - Azienda Ospedaliero-Universitaria Anna Meyer, Florence
  - Osp. dei Bambini V. Buzzi, ASST Fatebenefratelli Sacco, Milan
  - Azienda Ospedaliero-Universitaria di Parma Ospedale dei Bambini Pietro Barilla, Clinica Pediatrica, Parma
  - IRCCS Ospedale Pediatrico Bambino Gesù, Roma
- Poland (4):
  - MED-POLONIA Sp.z o.o., Poznan
  - Kliniczny Szpital Wojewodzki nr 2 im. Sw. Jadwigi Krolowej w Rzeszowie, Rzeszów
  - SPSK Nr 1 im. prof. Tadeusza Sokolowskiego PUM, Szczecin
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
- Romania (8):
  - Cen Med de Diagn si Trat Amb NEOMED, Brasov
  - Sana Monitoring, Bucharest
  - Medicover Hospitals, Bucharest
  - Institutul de Endocrinologie "C.I. Parhon", Bucharest
  - Spitalul Clinic Judetean de Urgenta "Sf. Apostol Andrei" Constanta, Constanța
  - Spitalul Clinic Judetean de Urgenta "Sf. Spiridon" Iasi, Iași
  - Spitalul Clinic Judetean Mures, Târgu Mureş
  - Spitalul Cl. de Urgenta pentru Copii Louis Turcanu Timisoara, Timișoara
- Serbia (3):
  - University children's clinic Belgrade - Department of Endocrinology, Belgrade
  - Clinical Center Nis - Clinic for Children's Internal Medicine, Niš
  - Institute for Child and Youth Health Care of Vojvodina - Endocrinology, Novi Sad
- Slovakia (3):
  - National Institute of Children's Diseases, Bratislava
  - Children's University Hospital Kosice, Košice
  - National Institute of Endocrinology and Diabetology, Ľubochňa
- Univerzitetni Klinicni Center Ljubljana - Pediatrics, Ljubljana, Slovenia
- Turkey (Türkiye) (4):
  - Ankara University, Faculty of Medicine, Ankara
  - Antalya Training and Research Hospital, Antalya
  - Kocaeli University Faculty of Medicine, Kocaeli
  - Karadeniz Technical University, Ortahisar